CLINICAL TRIAL: NCT06117514
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Dose-ascending Phase I Trial to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of Sudapyridine (WX-081) Tablets in Healthy Chinese Subjects
Brief Title: Sudapyridine (WX-081) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiatan Pharmatech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JYB0101
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — sudapyridine; Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Sudapyridine 30 mg single dose (Experimental): Participants received Sudapyridine 30 mg single dose orally.
  Interventions: Drug: Sudapyridine 30mg
- Sudapyridine 100 mg single dose (Experimental): Participants received Sudapyridine 100 mg single dose orally.
  Interventions: Drug: Sudapyridine 100mg SAD
- Sudapyridine 200 mg single dose (Experimental): Participants received Sudapyridine 200 mg single dose orally.
  Interventions: Drug: Sudapyridine 200mg SAD
- Sudapyridine 200 mg multiple doses (Experimental): Participants received Sudapyridine 200 mg orally for multiple doses.
  Interventions: Drug: Sudapyridine 200mg MAD
- Sudapyridine 300 mg multiple doses (Experimental): Participants received Sudapyridine 300 mg orally for multiple doses.
  Interventions: Drug: Sudapyridine 300mg MAD
- Placebo 100 mg single dose (Placebo Comparator): Participants received Placebo 100 mg single dose orally.
  Interventions: Other: Placebo tablet SAD
- Placebo 200 mg single dose (Placebo Comparator): Participants received Placebo 200 mg single dose orally.
  Interventions: Other: Placebo 200mg SAD
- Placebo 200 mg multiple doses (Placebo Comparator): articipants received Placebo 200 mg orally for multiple doses.
  Interventions: Other: Placebo tablet MAD
- Placebo 300mg multiple doses (Placebo Comparator): Participants received Placebo 300 mg orally for multiple doses.
  Interventions: Other: Placebo tablet MAD

INTERVENTIONS:
Drug: Sudapyridine 30mg — Sudapyridine capsule 30mg, orally, single dose
  Other Names: Sudapyridine capsule 30mg SAD
  Arms: Sudapyridine 30 mg single dose
Drug: Sudapyridine 100mg SAD — Sudapyridine tablet, 100mg orally, single dose
  Other Names: Sudapyridine tablet 100mg SAD
  Arms: Sudapyridine 100 mg single dose
Drug: Sudapyridine 200mg SAD — Sudapyridine tablet, 200mg orally, single dose
  Other Names: Sudapyridine tablet 200mg SAD
  Arms: Sudapyridine 200 mg single dose
Drug: Sudapyridine 200mg MAD — Sudapyridine tablet, 200mg orally once a day for 14 days
  Other Names: Sudapyridine tablet 200mg MAD
  Arms: Sudapyridine 200 mg multiple doses
Drug: Sudapyridine 300mg MAD — Sudapyridine tablet, 300mg orally once a day for 14 days
  Other Names: Sudapyridine tablet 300mg MAD
  Arms: Sudapyridine 300 mg multiple doses
Other: Placebo tablet SAD — Placebo tablet, 100mg orally, single dose
  Other Names: Placebo tablet 100mg
  Arms: Placebo 100 mg single dose
Other: Placebo 200mg SAD — Placebo tablet, 200mg orally, single dose
  Arms: Placebo 200 mg single dose
Other: Placebo tablet MAD — Placebo tablet, 200mg orally once a day for 14 days
  Other Names: Placebo tablet 200mg MAD
  Arms: Placebo 200 mg multiple doses
Other: Placebo tablet MAD — Placebo tablet, 300mg orally once a day for 14 days
  Other Names: Placebo tablet 300mg MAD
  Arms: Placebo 300mg multiple doses

SUMMARY:
The objective of this study is to evaluate the safety, tolerability as well as pharmacokinetics of Sudapyridine (WX-081) in Chinese volunteers.

DETAILED DESCRIPTION:
In this study, a single-center, randomized, double-blind, placebo-controlled, dose-ascending design was used to evaluate the safety, tolerability and pharmacokinetic characteristics of Sudapyridine (WX-081) tablets in healthy Chinese subjects using placebo as control.

This study was divided into two stages. The first stage evaluated the tolerance of single administration, pharmacokinetic characteristics, and the effect of food on PK. The second stage evaluated the tolerance of multiple administration and PK characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Weight: ≥50 kg; 19≤ body mass index (BMI) < 26 kg/m2;
* Considered healthy by the investigator based on a detailed history, thorough physical examination, clinical laboratory examination, 12-lead ECG, and vital signs results;
* No parenting plan and reliable contraception during the trial period and within 3 months after the last dose.

Exclusion Criteria:

* Allergic to any drug of the same category or its ingredients;
* A history of alcohol dependence or drug abuse;
* Laboratory obvious abnormalities;
* CYP3A4 potent inducer or inhibitor had been taken within 30 days prior to enrollment;
* Any serious cardiovascular, kidney, liver, blood, tumor, endocrine and metabolic, autoimmune or rheumatic diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of Sudapyridine | 0,1,2,3,4,6,8,12,24,48,72,96,120,144 hours post-dose
  PK parameter
Time to reach plasma Cmax (Tmax) of Sudapyridine | 0,1,2,3,4,6,8,12,24,48,72,96,120,144 hours post-dose
  PK parameter
Area under the plasma concentration-time curve (AUC) of Sudapyridine | 0,1,2,3,4,6,8,12,24,48,72,96,120,144 hours post-dose
  PK parameter
Terminal elimination half-life (t½) of Sudapyridine | 0,1,2,3,4,6,8,12,24,48,72,96,120,144 hours post-dose
  PK parameter
Volume of distribution (Vd/F) of Sudapyridine | 0,1,2,3,4,6,8,12,24,48,72,96,120,144 hours post-dose
  PK parameter
Apparent clearance (CL/F) of Sudapyridine | 0,1,2,3,4,6,8,12,24,48,72,96,120,144 hours post-dose
  PK parameter
Elimination rate constant Ke of Sudapyridine | 0,1,2,3,4,6,8,12,24,48,72,96,120,144 hours post-dose
  PK parameter
Number of participants with adverse events (AEs) or Serious Adverse Events (SAEs) | 0,1,2,3,4,6,8,12,24,48,72,96,120,144 hours post-dose
  safety parameter

CONTACTS AND LOCATIONS:
Overall Officials: Yun Liu, Principal Investigator — Shanghai Xuhui District Central Hospital
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No